CLINICAL TRIAL: NCT06063005
Title: Clinical Study of Translocated Internal Limiting Membrane Flap Reposition for the Treatment of Idiopathic Macular Hole
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government)
Responsible Party: Principal Investigator, Peiquan Zhao, Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-22-084
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Translocation (Experimental)
  Interventions: Procedure: Translocation ILM Flap
- Peeling (Active Comparator)
  Interventions: Procedure: ILM Peeling

INTERVENTIONS:
Procedure: Translocation ILM Flap — After vitrectomy, the ILM was dissected from the macula to the vascular arch, and the retina in the fissure area was fully released to make an MH-centered, approximately 2DD-square, ILM flap with a tip (approximately 500μm wide) above; the ILM flap was transposed approximately 25-30 degrees along the tip to the inferior temporal area with the assistance of heavy water, and a total of 1ml of perfluorodecalin fluid (heavy water) was injected to cover the MH area with the ILM flap, and the original ILM defect area corresponding to the MH was transposed to the outside of the MH. The heavy water is replaced by liquid/gas exchange. Ophthalmic 13% perfluoropropane gas (AL.CHI.MI.A. Srl) was chosen as the postoperative intraocular filling.
  Arms: Translocation
Procedure: ILM Peeling — After vitrectomy, internal limiting membrane peeling up to the vascular arcade, thorough loosening of the macular hole area of the retina, and fluid/gas exchange. An eye-specific 13% perfluoropropane gas (AL.CHI.MI.A. Srl) was chosen for intraocular tamponade after the operation.
  Arms: Peeling

SUMMARY:
The main objective of this study is to evaluate the therapeutic effectiveness of the internal limiting membrane (ILM) peeling and translocation surgery compared to the conventional surgical approach for treating large idiopathic macular hole (IMH) through a well-designed prospective randomized controlled clinical trial. This study aims to compare the new surgical approach to the conventional approach in terms of improving visual function, promoting macular retinal anatomical healing, and enhancing patients' quality of life. By conducting this prospective clinical trial, establishing a database, and generating clinical reports and evidence-based medicine on the therapeutic efficacy of the ILM peeling and translocation surgery for large IMH.

ELIGIBILITY:
Inclusion Criteria:

* Participants who can understand the purpose of this clinical trial, volunteer to participate, sign an informed consent form, and can complete the postoperative follow-up on time.
* Participants diagnosed with idiopathic macular hole (IMH).
* Based on OCT scans, the minimum horizontal diameter of the macular hole is >500 and <900 µm.
* Participants with an axial length <26.0mm and a myopic degree lower than 6D.
* For participants with bilateral macular holes, the eye with a larger hole diameter will be included.

Exclusion Criteria:

* Patients with the following retinal disorders: age-related macular degeneration, epi-macular membrane neovascularization, non-macular retinal tears, lesions of the retinal pigment epithelium and choroid, inherited or degenerative retinal diseases, optic neuropathies, retinal vascular diseases; patients with large macular holes accompanied by retinal detachment;
* Patients with high myopia (axial length ≥ 26.0mm and myopia exceeding 6D);
* Patients with a history of ocular trauma or retinal laser treatment;
* Patients with glaucoma, ocular infections, inflammations, tumors, corneal diseases, or amblyopia;
* Patients with contraindications to vitrectomy;
* Patients with severe or unstable systemic diseases;
* Patients with a fasting blood glucose level ≥ 9mmol/L before surgery;
* Patients who participated in other clinical trials involving drugs or medical devices within 30 days prior to screening;
* Patients with a history of intraocular surgery within 3 months prior to screening;
* Patients with reduced visual function or vision in the contralateral eye as determined by the investigator;
* Patients who are not considered suitable for enrollment by the investigator for other reasons.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | 1 week, 1 month, 3 months, 1 years, 2 years after the operation
  The best corrected visual acuity indicates the best visual acuity with proper refractive correction.

SECONDARY OUTCOMES:
Closure rate | 1 week, 1 month, 3 months, 1 years, 2 years after the operation
  MH closure is mainly reflected in the outer layer of continuity closure shown on OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Peiquan Zhao, Dr., Study Chair — Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine Shanghai
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No